CLINICAL TRIAL: NCT03899675
Title: Impact of Caffeine Intake Before Exercise on the Neural Regulation of the Cardiovascular System in Physically Active Adults
Brief Title: Impact of Caffeine Intake on Autonomic Parameters in the Exercise of Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pernambuco (Other)
Responsible Party: Principal Investigator, Cicero Jonas Rodrigues Benjamim, Principal Investigator, University of Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UPernambuco
Record Dates: First submitted 2019-03-26; First posted 2019-04-02 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Autonomic Nervous System; Cardiovascular Outcomes
Keywords: Caffeine; Exercise; Heart Rate Variability; Autonomic Nervous System; Cardiovascular Risk Factor
MeSH Terms: conditions — Motor Activity | interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: It is a randomized, single-blind clinical trial
Who Masked: Participant
Masking Description: The research will be divided into two moments, in which subjects will participate in the same experiment on two different and non sequential days, and on the first day, the measurement of data will occur without the ingestion of caffeine or placebo. Participants will be randomized at the end of the first evaluation.
  The randomization of the volunteers to define the groups will be performed using random numbers obtained at www.randomized.com. Subjects will be allocated to one of two groups: I) strength training and caffeine; II): strength training and placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caffeine (Experimental): Volunteers will ingest 300mg caffeine one hour before strength training.
  Interventions: Other: Caffeine
- Placebo (Placebo Comparator): Volunteers will ingest 300mg placebo one hour before strength training.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — On the first day of collection, the volunteers will not take placebo intake, the data will be collected in a standardized way, respecting the times defined for the analysis of the cardiac activity. Then the collection will be continued. On the next day of evaluation, volunteers will receive a capsule containing 300 mg of placebo and will be advised to consume 1 hour before the procedure.
  Arms: Placebo
Other: Caffeine — On the first day of collection, the volunteers will not take caffeine intake, the data will be collected in a standardized way, respecting the times defined for the analysis of the cardiac activity. Then the collection will be continued. On the next day of evaluation, volunteers will receive a capsule containing 300 mg of caffeine and will be advised to consume 1 hour before the procedure.
  Arms: Caffeine

SUMMARY:
The objective of this study was to evaluate the variability of the heart rate of exercise physicists with and without caffeine intake. Practitioners of resisted physical exercise, specifically bodybuilding, who are young adults between the ages of 18 and 30 will participate in the study. To define the sample size, a sample calculation was performed based considering as variable the RMSSD index (square root of the square mean of the differences between the adjacent normal iRRs). The significant difference magnitude assumed was 12 ms, considering a standard deviation of 16.2 ms, with alpha risk of 5% and beta of 80%. A minimum of 14 subjects per group were required in the survey. A total of 32 subjects will participate in the research, being these divided and allocated in different groups. Sampling will be of the intentional kind.

DETAILED DESCRIPTION:
Caffeine supplementation has been studied in several sports modalities with the objective of investigating its repercussions on athletes' physical performance. Caffeine may lead to an obstruction of adenosine receptors (A1 and A2) and increase the activity of the Autonomic Nervous System (ANS) by releasing catecholamines in plasma, inducing tachycardia and elevating blood pressure. Such modulation of nervous system activity can be traced by assessing heart rate variability (HRV). HRV is one of the most practical methods to analyze the physiological functioning of ANS, both in pathological conditions of the individual and in the induction of other variables, being a noninvasive measure of cardiac autonomic modulation markers that analyzes the peak-R intervals a peak-R (RRI) of consecutive heartbeat. The objective of this study was to evaluate the variability of the heart rate of exercise physicists with and without caffeine intake. Practitioners of resisted physical exercise, specifically bodybuilding, who are young adults between the ages of 18 and 30 will participate in the study. To define the sample size, a sample calculation was performed based considering as variable the RMSSD index (square root of the square mean of the differences between the adjacent normal iRRs). The significant difference magnitude assumed was 12 ms, considering a standard deviation of 16.2 ms, with alpha risk of 5% and beta of 80%. A minimum of 14 subjects per group were required in the survey. A total of 32 subjects will participate in the research, being these divided and allocated in different groups. Sampling will be of the intentional kind.

The expected benefits with the result of this research are to instigate the creation of new lines of research in this context, being able to intervene in a more effective way in practitioners of physical exercise of strength, with the possibility of prevention to the autonomic alterations that are associated with the consumption of stimulant supplements, such as caffeine, and its consequences on the cardiovascular system.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18 to 30 years of age
* Body Mass Index (BMI) within the range of Eutrophy (18.5 to 24.9kg / m²)
* Experience with resistance training, uninterrupted for at least 3 months and weekly frequency of 3 sessions or more
* Do not use any medication that may interfere with cardiac autonomic modulation
* Do have no skeletal muscle damage.

Exclusion Criteria:

* Smoking patients
* As well as individuals who have already used anabolic steroids
* Cardiorespiratory diseases
* Cardiometabolic diseases
* Neurological disorders
* Other known compromises that prevent the subject from performing the procedures.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Caffeine effects on heart rate variability (based on frequency, time domain and Chaos) | up to 1 year
Blood pressure (mmHg) | up to 1 year
  Caffeine effects blood pressure recovery following strength exercise
Heart rate (beats per minute) | up to 1 year
  Caffeine effects heart rate recovery following strength exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Cicero Jonas Rodrigues Benjamim, Juazeiro do Norte, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No
No, we intend to disseminate the results in scientific journals.